CLINICAL TRIAL: NCT02881268
Title: Study of Immunosuppression Biomarkers Acquired in Patients Hospitalized in Intensive Care Unit
Acronym: IMPRIM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_9903_IMPRIM
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Patient Hospitalized in Intensive Care Unit
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient with sepsis: Patient hospitalized in intensive care unit
  Interventions: Other: blood sample
- Patient without sepsis: Patient hospitalized in intensive care unit
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Open-label, non-randomized, prospective, single center, observational, translational study

DETAILED DESCRIPTION:
The aim of this trial is to study immunosuppression biomarkers in patients hospitalized in intensive care unit in comparison to non-septic patients.

Prevalence of immunosuppression acquired in intensive care unit will be studied and patients most likely to develop nosocomial infection will be early identified

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient hospitalized in intensive care unit for any reason
* Patient with infection started less than 5 days before admission
* Patient with mechanical ventilation or not
* Patient with arterial catheter for an invasive monitoring of blood pressure
* Patient informed about the study protocol and approved to participate.
* Patients hospitalized for a severe bacterial infection (severe sepsis or septic shock)
* Patient hospitalized for a non-infectious disease

Exclusion Criteria:

* Pregnancy
* Advanced immunosuppression defined by proved humoral or cellular impairment by continuous administration of steroids at any dose since more than one month before hospitalization, transplantation, radiotherapy or chemotherapy in the preceding year
* Initiation of an immunosuppressive therapy as chemotherapy, cyclophosphamide or high dose corticotherapy (>0.5mg/kg/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in intensive care unit with or without sepsis
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Detection of immunosuppression biomarkers in septic and non-septic patients hospitalized in intensive care unit | Day 14

SECONDARY OUTCOMES:
Association of immunosuppression biomarkers with occurrence of events reflecting a clinical immunosuppression | Day 14
  Study of CMV reactivation and nosocomial infections
Association of immunosuppression biomarkers with patients demographic data | Day 14
  Record of patient age and gender
Association of immunosuppression biomarkers with patients clinical data | Day 14
  Record of severity score, duration of hospitalization, duration of mechanical ventilation, morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No